CLINICAL TRIAL: NCT02837172
Title: Diagnosis of Parkinson's Disease and Prediction of Progression Using Diffusion Weighted Imaging
Brief Title: Diagnosis of PD and PD Progression Using DWI
Acronym: K23
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dr. Frank Michael Skidmore, Assistant Professor of Neurology, University of Alabama at Birmingham
Other Study IDs: K23NS083620 (NIH)
Record Dates: First submitted 2016-04-29; First posted 2016-07-19 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Parkinson's disease from UAB: MDS-UPDRS,Montreal Cognitive Assessment, PDQ-39, Diffusion Weighted Imaging (DWI), and neurological examination.
  Interventions: Other: Diffusion Weighted Imaging (DWI)
- Parkinson's disease from PPMI dataset: Obtain retrospective and prospective de-identified data from the The Parkinson's Progression Markers Initiative (PPMI) dataset on Parkinson's disease (PD) subjects that have the following characteristics: within 2 years of diagnosis, positive DaTscan, and not (at study entry) on any PD related medication.
- Controls from PPMI dataset: Obtain retrospective and prospective de-identified DTI imaging and data from the PPMI dataset

INTERVENTIONS:
Other: Diffusion Weighted Imaging (DWI) — MDS-UPDRS,Montreal Cognitive Assessment, PDQ-39, DTI imaging (MRI), and neurological examination.
  Expert evaluation: Record review, PD Medical History and PD Family History Form, the Montreal Cognitive Assessment, PDQ-39. standard, full, neurological examination, and MDS-UPDRS
  Groups: Parkinson's disease from UAB

SUMMARY:
This project will evaluate the utility of diffusion tensor imaging (DTI) as an adjunctive method to improve early diagnosis of Parkinson's disease (PD). Two populations will be evaluated in this study: 1) Individuals with uncertain PD diagnosis who receive a DaTscan, and 2) individuals with well characterized PD and healthy controls, drawn from the fully enrolled Parkinson's Progression Markers Initiative (PPMI) PD and control cohorts.

DETAILED DESCRIPTION:
Specific Aim 1a: Compare the outcome of a DTI based prediction with a contemporaneous clinical DAT scan in 100 subjects with suspected parkinsonism, and determine rate of concordance between the two diagnostic techniques.

Specific Aim 1b: Compare predictive accuracy of a baseline DTI with a "gold standard" expert diagnosis after 36 months of follow up in 100 subjects receiving DaTscan for suspected parkinsonism.

Specific Aim 2a: Use TBM to evaluate volume and cross-sectional caliber (based on point-wise fiber track direction) of the fimbria, pallidonigral tracts, and subthalamic-nigral tracts in PD and healthy controls. Ascertain if changes in white matter volume and caliber can be used to predict presence of PD from the PPMI study. Secondarily, using a model free approach, determine what white matter features based on TBM predict presence of disease.

Specific Aim 2b: Use TBM to determine if an increased rate of change in volume and cross-sectional caliber of the fimbria, and hypertrophic pallidonigral, and subthalamic-nigral tracts identified in aim 2a, are associated with a more rapid rate of disease progression in PD. Secondarily, using a model free approach, determine what white matter features based on TBM predict a faster rate of disease progression over the 5 year course of the PPMI study.

Specific Aim 3a: Compare DTI FA in TD-PD and PIGD-PD in the thalamus and lobule IX of the cerebellum , studying subjects from the PPMI study. Predict signal in these regions will predict phenotypic expression of disease. Using TBM and bootstrapping, determine the relationship between phenotypic expression of disease and white matter input/output pathways from the thalamus, and from lobule IX of the cerebellum.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 and older
* Referred for clinical DaTscan for possible PD
* Controls from the PPMI dataset.

Exclusion Criteria:

* Pregnant women
* Participants that cannot participate in MRI (metallic artifact or other contraindication(s) to MRI at 3T)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 PD subjects with DaTscan, and 210 (140 PD/70 control) from the PPMI dataset
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
MRI and DAT scan: Accuracy of diagnosis of Parkinson's disease in a clinically relevant population | 3-5 years
  The study investigators will measure if MRI, specifically diffusion weighted imaging, can predict existence of Parkinson's disease. The study investigators will valuate if the derived MRI prediction matches or exceeds the accuracy of DATscan in detecting Parkinson's disease. The clinical/radiology reading of the DAT scan will determine the DAT scan diagnosis. The MRI scan diagnosis will be derived from statistical analysis of the full 5-dimensional brain DWI signal, as well as signals such as MRI T1 and resting fMRI signal. Methods of analysis will include using standard statistical techniques, the investigators published novel statistical techniques, and techniques such as Deep Learning and other artificial intelligence/learning algorithms.

SECONDARY OUTCOMES:
Can MRI profile risk for tremor and postural instability in PD | 3-5 years
  The study investigators will measure if MRI, specifically diffusion weighted imaging, can predict at disease onset which individuals with Parkinson's disease are at risk of developing significant postural instability and gait dysfunction.The MRI scan prediction will be derived from statistical analysis of the full 5-dimensional brain DWI signal, as well as signals such as MRI T1 and resting fMRI signal. Methods of analysis will include using standard statistical techniques, the investigators published novel statistical techniques, and techniques such as Deep Learning and other artificial intelligence/learning algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Skidmore, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
progress report information to NIH